CLINICAL TRIAL: NCT03405298
Title: Reducing Inappropriate Benzodiazepine Use Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Donovan Maust, Professor of Psychiatry, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00133623; 20180230-00 (Other Grant/Funding Number: Michigan, State of, Health and Human Services, Department of Health and Human Services)
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Long Term Use of Benzodiazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Material with Collaborative Care available (Active Comparator): In addition to the material described below, these patients are seen in clinics with behavioral health collaborative care (BHCC), which includes a care manager in the primary care provider's office along with a consulting psychiatrist. If a patient receives the brochure and would like to taper their benzodiazepine, their provider can refer them to the BHCC care manager who can provide education and anxiety and insomnia self-management strategies, while the BHCC psychiatrist will make recommendations regarding the medication taper back to the primary care provider.
  Interventions: Behavioral: Educational Material; Behavioral: Supplemental Collaborative Care
- Educational Material Only (Active Comparator): Patients will receive an 8-page educational brochure that presents information about potential harms of these medications and a vignette about a patient that successfully stopped. It does NOT suggest patients to stop on their own, but rather suggests they speak with their provider.
  Interventions: Behavioral: Educational Material

INTERVENTIONS:
Behavioral: Educational Material — Educational material is in the form of a brochure
Behavioral: Supplemental Collaborative Care — Supplemental care management consist of meeting with a behavioral health care manager over five sessions in-person or via phone call; the care manager will review patient information with the consulting psychiatrist, who can then make recommendations back to the primary care provider
  Arms: Educational Material with Collaborative Care available

SUMMARY:
The goal of this project is to reduce chronic benzodiazepine use through two approaches: direct patient education or direct patient education paired with additional support and encouragement from a behavioral health care manager.

DETAILED DESCRIPTION:
This is a State of Michigan/Medicaid Match project proposal. These proposed projects are developed to address specific goals for Medicaid policies, procedures, and model programs for Medicaid Recipients in Michigan.

Benzodiazepine use in the United States is common and increases with age, used by 8.7% of patients aged 65-80 years. Benzodiazepines-which include well-known medications such as Xanax, Ativan, and Klonopin-are most commonly used for anxiety and insomnia, even though psychotherapy and alternative medications are now recommended preferentially over benzodiazepines. Use is a particular concern among older adults, given the links between benzodiazepine prescribing and a variety of adverse outcomes including falls, fractures and motor vehicle accidents.

Attempts to reduce benzodiazepine use have met with limited success in the real world, as patients are reluctant to consider the possibility of stopping them and providers are reluctant to even suggest the possibility. In the course of a brief return visit in primary care, providers simply do not have the time or incentive to engage in a potentially difficult, lengthy discussion with patients about reducing or stopping their benzodiazepine.

The goal of this project is to evaluate direct patient education compared to direct patient education paired with additional support and encouragement from a care manager in order to reduce chronic benzodiazepine use. Strategies to help reduce benzodiazepine use are of great interest to providers and our findings would have significance for all providers, and may even conceivably improve the care of patient both inside and outside the Medicaid program.

ELIGIBILITY:
Inclusion Criteria:

* With a prescription BZD supply covering ≥20% of days in the preceding 12 months ("chronic").

Exclusion Criteria:

* Patients with BZD supply <20% days in past 12 months
* Patients with ICD-10 codes for dementia (derived from encounter diagnosis codes)
* long-term care residents (ICD-10 codes Z59.3 and Y92.199)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Change in avg. daily dose of benzodiazepine prescribed in lorazepam-equivalent mg | 3 months
  Compare the average daily dose during month 3 to the baseline average daily dose
Change in avg. daily dose of benzodiazepine prescribed in lorazepam-equivalent mg | 6 months
  Compare the average daily dose during month 6 to the baseline average daily dose

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) | 3 months
  The PHQ-8 is a self-report instrument assessing 8 DSM-IV symptoms of depression, this measure will be conducted at 3 months, with total scores ranging from 0 (low) to 24 (high); scores ≥10 suggest the presence of Major Depressive Disorder.
Generalized Anxiety Disorder 7-Item Scale (GAD-7) | 3 months
  The GAD-7 total score ranges from 0 (low) to 21 (high), with "cut scores" for mild (5), moderate (10), and severe anxiety (15); will be conducted at 3 months.
Insomnia Severity Index (ISI) | 3 months
  ISI is a valid and sensitive measure to detect changes in perceived sleep difficulties, ranging from 0-28. Scores of 0-7 are categorized as no clinically significant insomnia, 8-14 subthreshold insomnia, 15-21 clinical insomnia (moderate severity), 22-28 clinical insomnia (severe).
Alcohol Use Disorders Identification Test (AUDIT-C) | 3 months
  Hazardous Alcohol Use will be assessed using the AUDIT-C which assesses average alcohol consumption (quantity and frequency) and binge drinking (6 or more) over the past 3 months on a scale of 0 (none) to 12 (heavy alcohol use).The cut-off scores for hazardous drinking are 3 for women and 4 for men.
PHQ-8 | 6 months
  The PHQ-8 is a self-report instrument assessing 8 DSM-IV symptoms of depression, this measure will be conducted at 6 months, with total scores ranging from 0 (low) to 24 (high); scores ≥10 suggest the presence of Major Depressive Disorder.
GAD-7 | 6 months
  The GAD-7 total score ranges from 0 (low) to 21 (high), with "cut scores" for mild (5), moderate (10), and severe anxiety (15).
ISI | 6 months
  ISI is a valid and sensitive measure to detect changes in perceived sleep difficulties, ranging from 0-28. Scores of 0-7 are categorized as no clinically significant insomnia, 8-14 subthreshold insomnia, 15-21 clinical insomnia (moderate severity), 22-28 clinical insomnia (severe).
AUDIT-C | 6 months
  Hazardous Alcohol Use will be assessed using the AUDIT-C which assesses average alcohol consumption (quantity and frequency) and binge drinking (6 or more), this measure will be conducted at 6 months, on a scale of 0 (none) to 12 (heavy alcohol use).The cut-off scores for hazardous drinking are 3 for women and 4 for men.

CONTACTS AND LOCATIONS:
Overall Officials: Donovan Maust, MS, MD, Principal Investigator — University of Michigan
Locations (1):
- Department of Psychiatry, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No